CLINICAL TRIAL: NCT04960683
Title: The Effectiveness of Robotic Assisted Gait Training as an Adjunct to Traditional Physiotherapy in Cerebral Palsy
Acronym: RAGT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatima College of Health Sciences (Other)
Responsible Party: Principal Investigator, Dragana Djuric, Instructor in physiotherapy, Fatima College of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INTSTF018PHY20
Record Dates: First submitted 2021-01-13; First posted 2021-07-14 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Cerebral Palsy
Keywords: Children; Lokomat
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic -assisted gait training group using Lokomat device (Experimental): * 5 sessions of 40 minutes of conventional therapy and
  * 5 sessions of 40 minutes on Lokomat per week
  Interventions: Device: Lokomat training
- Traditional therapy group (Active Comparator): • 5 sessions of 40 minutes of conventional therapy
  Interventions: Device: Lokomat training

INTERVENTIONS:
Device: Lokomat training — Control group will receive the routine conventional physiotherapy treatment and the treatment for this group consists of the following:
  Conventional therapy protocol:
  * 5 sessions of 45 minutes a week, each session includes:
  * 5 minutes of stretching exercise
  * 20 minutes of strengthening exercise
  * 10 minutes of balance exercise
  * 10 minutes of gait training
  Experimental group will receive 45 min of Lokomat in addition to the conventional approach (as explained above). Since Lokomat appointments can be only 8 per day, it is planned to have two groups of 8 participants for 4 weeks each. The Lokomat training include the following:
  * 5 sessions of 45 minutes of conventional therapy (same as above) per week
  * 5 sessions of 45 minutes on Lokomat per week
  Other Names: Conventional therapy

SUMMARY:
Need for study

There are a few studies published on this topic from various parts of the globe and the results are mixed. Hence further research is required in this area and none of the studies have included samples from the Middle East.

Some studies done in this area focus on biomechanical aspects of gait (Cherni, 2018) and our study mainly focuses on functional aspects of gait and quality of life.

Studies done on this area focus highly on gait components and very little is available on the literature on improving balance. Since balance and stability are crucial for walking, it was decided to exclusively assess balance.

Due to a wide range of therapeutic benefits, it is paramount to evaluate the effectiveness of different therapies provided to improve gait.

Aim of the study:

The aim of the proposed research is to investigate the effectiveness of robotic assisted gait training using Lokomat device as an adjunct in improving gait, balance and quality of life in children with cerebral palsy.

DETAILED DESCRIPTION:
Background: Gait and balance have been a major issue faced by cerebral palsy children. Cerebral Palsy is the most common condition affecting around 2-2.5 children of 1000 live births (1 in every 400 children) over the last 20 years in the Western world (Levit, 2019). Cerebral Palsy causes complex issues related to physical, psychological and social functions. Active participation and the highest level of independence during daily living are primary goals for cerebral palsy children (Aurich, 2015). One of the major problems that limits activities of daily living is relate to gait and balance in cerebral palsy. From the past one-decade, the popularity of robotic assisted gait training devices have been increasing. There are a studies published on this topic from various parts of the globe and the results are mixed. Recent publications have demonstrated robotic assisted gait training benefits people with cerebral palsy, specifically in increasing walking speed and endurance (Carvalho, 2017). However, the efficacy of robotic assisted gait training in improving gait and balance is not well researched. This study will be the first one in the United Arab Emirates studying the local population and mainly focusing on functional aspects of gait, balance and quality of life.

Aims: The main aim is to investigate the effectiveness of robotic -assisted gait training as an adjunct to traditional physiotherapy to improve gait, balance and quality of life in children with cerebral palsy.

Research hypothesis: Robotic -assisted gait training applied as adjunct to traditional therapy could improve balance, walking and quality of life in children with cerebral palsy.

Methodology: The participants attending the outpatient clinic at Zayed Higher Organization for People of Determination, Abu Dhabi will be invited to take part in the study. They will be randomly allocated to two groups. This study proposes to have 50 participants with at least 25 in each group. The participants will all have spastic form of cerebral palsy as possible with the age of 4-18 years. All the participants will have to have be at Gross Motor Function Classification Level (GMFCS) level I- IV. The robotic -assisted gait training include 5 sessions per week, of 40 min long session during one-month period. The conventional physiotherapy includes 5 sessions per week of 40 min long session during one-month period. The primary analysis will be the pre to post-test differences of the Gross Motor Function Measure (GMFM-88),dimension D & E, 10 meters walk test, 6 minute walk test, Pediatric Balance Scale, Cerebral palsy Quality of Life questionnaire between experimental and control group.

Data analysis: Data will be statistically analysed using one-way anova. Descriptive statistics and graphic displays will be present for all outcomes for interventions comparing robotic -assisted gait training with traditional physiotherapy training.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral palsy with spastic and mix form

  * Gross Motor Function Classification System (GMFCS from level II to IV)
  * Age 4 to 18
  * No contraindications for the training in the Lokomat
  * Able to follow simple instructions

Exclusion Criteria:

* On botox injection within the last 6 months (as the effect of botox wear out in 6 months)

  * Surgery within the last one year
  * Fixed contractures and/or with bone instability
  * Baclofen infusion pumps in situ
  * Seizure disorder that is not controlled by medication (if on medication, must not have had a seizure in the last 12 months);
  * Open skin lesions or vascular disorder of lower extremities;
  * Having participated in another Lokomat training regime within the previous 3months as well as a change in concomitant treatment within the last 4 weeks before or during the study period

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2020-11-08 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure ( GMFM- 88) - dimension D & dimension E | Baseline time 0 and up to 8 weeks
  This is the validated test designed to measure change in gross motor function over time in children with cerebral palsy. Dimension D consist of 13 items for standing ability and dimension E has 24 items to assess walking, jumping and running in cerebral palsy children. Its a four point scoring system. Specific descriptors for each score is given in the Manual of GMFM-88.
6 minute Walk test | Baseline time 0 and up to 8 weeks
  The test has been selected as a measure of gait endurance. This is validated test requiring individuals to walk 6 minutes on flat hard floor. Scoring is walking distance.
10 meters Walk test | Baseline time 0 and up to 8 weeks
  The test has been selected as a measure of gait speed. This is validated test requiring individuals to walk on flat hard floor at their comfortable speed for 10 meters.
Pediatric Balance Scale | Baseline time 0 and up to 8 weeks
  14 items valid scale is used to assess functional balance skills in children with spastic cerebral palsy.
Cerebral Palsy Quality of Life questionnaire for child (CP QOL-child) and Cerebral Palsy Quality of Life questionnaire for adolescent (CP QOL- teen) | Baseline time 0 and up to 8 weeks
  This Arabic validated CP QOL- child for age 4-12 and CP QOL- teen for age 13-18 questionnaires are used in the parent version. Its assesses 7 domains on a 9 level point Likert scale.

SECONDARY OUTCOMES:
Range of motion | Baseline time 0 and up to 8 weeks
  Measuring range of motion in hip, knee, ankle joint using the reliable tool called goniometer.
The Oxford scale | Baseline time 0 and up to 8 weeks
  The most commonly used scale for testing muscle strength.
Modified Ashworth Scale | Baseline time 0 and up to 8 weeks
  It is a muscle tone assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Dragana Djuric, Principal Investigator — FCHS
Locations (1):
- Fatima College of Health Sciences, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No